CLINICAL TRIAL: NCT06283433
Title: A Dried Blood Spot Sampling Method for Vancomycin and Creatinine Monitoring: Effectiveness Demonstrated in Outpatient Parenteral Antibiotic Therapy Service
Brief Title: A Dried Blood Spot Sampling Method for Vancomycin and Creatinine Monitoring for OPAT
Acronym: ADVANCEDOPAT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Birgit Koch, Professor, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: NL83813.078.23
Record Dates: First submitted 2023-10-30; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Infection, Bacterial
Keywords: microsampling; vancomycin; creatinine; dried blood spot
MeSH Terms: conditions — Bacterial Infections | interventions — Phlebotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (venipuncture) (Active Comparator): Conventional blood sampling via venipuncture method by a skilled drawing facility
  Interventions: Diagnostic Test: Venipuncture
- Intervention Group (DBS) (Experimental): Blood sampling via dried blood spotting (DBS) method at patient's home
  Interventions: Diagnostic Test: Finger Prick

INTERVENTIONS:
Diagnostic Test: Finger Prick — Blood sample obtained via drop of capillary blood by finger prick onto filter paper
  Other Names: Dried Blood Spot Sampling
  Arms: Intervention Group (DBS)
Diagnostic Test: Venipuncture — Blood sample obtained trough venipuncture
  Arms: Control Group (venipuncture)

SUMMARY:
The Outpatient Parenteral Antibiotic Therapy (OPAT) service consists of providing antimicrobial therapy through parenteral infusion without hospitalization. This service is provided to stable patients otherwise ready for hospital discharge. Generally, the clinical monitoring for this patient population is minimal. However, clinical monitoring of vancomycin, an antibiotic widely used during OPAT, can be intensive primarily due to therapeutic drug monitoring. To ensure optimal treatment and minimize nephrotoxicity and microbial resistance, TDM and monitoring of serum creatinine levels are crucial during vancomycin therapy. TDM of vancomycin with OPAT presents a challenge for patients who must frequently travel to blood sampling facilities or the hospital for measurements. An alternative sampling method for TDM is the dried blood spot (DBS) method, which involves collecting a small drop of capillary blood from a finger prick onto filter paper. By implementing the DBS sampling method, the amount of outpatient visits regarding vancomycin treatment in OPAT can be reduced. Furthermore, the addition of measuring a biochemical parameter, such as renal function with serum creatinine, could lead to even less outpatient visits during OPAT. To date, studies investigating the effectiveness of DBS sampling of vancomycin and creatinine in terms of reducing outpatient visits have not yet been conducted in the OPAT population.

DETAILED DESCRIPTION:
The use of vancomycin in OPAT services is widespread, however a drawback of its use is the need for laboratory monitoring of the vancomycin concentration which requires patients to travel to a blood sampling facility or the hospital for blood sampling. At most hospitals at least one or two blood samples per week are obtained for vancomycin drug monitoring from a patient in OPAT service receiving vancomycin. Conventional blood sampling involves an invasive procedure of drawing blood from a vene through a venipuncture, this is performed by a qualified health care worker at a blood drawing facility (often performed by a nurse in the hospital). Besides the burden for the patient to travel to a blood sampling facility the costs also have to be taken into account, contributing to a higher cost for OPAT services.

The hospital pharmacy laboratory of Erasmus University Medical Center has developed and clinically validated a dried blood spot (DBS) assay for measuring vancomycin and creatinine (ADVANCED study). The use of dried blood spot collection to quantify drug concentrations is an innovative technique that requires only a simple finger prick instead of an invasive venipuncture. Consequently, this is less painful and stressful for the patient than conventional blood sampling. DBS can be performed by taking a low-volume finger prick samples (10 to 20 μl) on filter paper. Finger samples can be taken and stored with a desiccant, without the need for processing and freezing of plasma. A small-diameter disc, or chad, can be subsequently punched out from the filter paper, and the drug can be eluted into a liquid matrix prior to a liquid chromatography-mass spectrometry (LC-MS) assay. The main benefit of DBS sampling is that it allows for the ease of self-sampling at home. DBS offers several other practical advantages over conventional plasma sampling. These advantages include lower sample volume requirements, simplified collection techniques, and less restrictive transport and storage conditions.

DBS sampling eliminates the need to travel to a sampling facility as no healthcare professionals are involved in the sampling process. To date, studies investigating the effectiveness of DBS sampling in terms of reducing outpatient visits have not been conducted in the OPAT population. OPAT is provided for patients who are stable and healthy enough to leave the hospital and clinical monitoring of these patient population is minimal. However, clinical monitoring of vancomycin therapy during OPAT is intensive due to TDM of vancomycin. Most protocols oblige at least once weekly TDM of vancomycin, which contributes to outpatient visits. By implementing DBS sampling the investigators hypothesize that the number of outpatient visits regarding vancomycin therapy in OPAT services can be reduced. Furthermore, this effectiveness may increase when a biochemical parameter such as renal function parameter (i.e. creatinine) are measured along with drug concentrations (leading to even less outpatient visits); the benefit of this has not been investigated yet.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 and over
* Able to understand written information and able to give informed consent
* Hospitalized
* Treated with intravenous vancomycin and to be discharged with vancomycin OPAT service with minimal 1 planned outpatient vancomycin TDM order
* Able and willing to perform finger pricks for dried blood spot sampling, or able and willing to undergo finger pricks performed by family members or other caregivers
* Able and willing to fill in questionnaires

Exclusion Criteria:

* Former participation in this trial
* Cognitive dysfunction or other dysfunctionalities which makes the patient unable to draw blood by a finger prick or fill out questionnaires
* Unable to sample an adequate DBS after training in the hospital (this is also applicable for family members or other caregivers who are failing to perform adequate DBS sampling for the patient)

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2023-10-25 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
To compare the number of outpatient visits in the control group versus the intervention group at day 28 | 28 days after discharge
  Number of outpatient visits

SECONDARY OUTCOMES:
Outcomes regarding outpatient visit | 28 days after discharge
  * To compare the number of outpatient visits with the sole purpose of vancomycin TDM in the control group versus intervention group (phlebotomy visits)
  * To compare the number of outpatient visits with the sole purpose of laboratory sampling (with and without TDM) in the control group versus intervention group
  * To compare the number of outpatient visits regarding vancomycin therapy without laboratory sampling in the control group versus intervention group
  * To compare the number of outpatient visits regarding vancomycin therapy including laboratory sampling (with and without TDM) in the control group versus intervention group
  * To compare the number of vancomycin therapy related telephone consultations in the control group versus intervention group
Sampling outcomes | 28 days after discharge
  - To compare the number of correct blood sampling in the control group versus intervention group
Satisfaction with blood sampling based on the theoretical framework of acceptability questionnaire (TFA) | 28 days after discharge
  - To investigate if dried blood spot sampling of vancomycin leads to a higher patient satisfaction score (questionnaire) compared with conventional sampling in OPAT service. A higher score means a higher patient satisfaction (maximum score is 7)
Cost outcomes | 28 days after discharge
  * To compare patient costs in the control group versus intervention group
  * To compare costs related to loss of productivity in the control group versus intervention group
  * To compare health care costs in the control group versus intervention group
  * To compare societal costs (total of all costs) in the control group versus intervention group
Clinical outcomes | 28 days after discharge
  - To compare clinical outcomes in the control group versus intervention group
TDM outcomes | 28 days after discharge
  To compare the relative number of vancomycin measurements in the control group versus intervention group
Logistical outcomes | 28 days after discharge
  To compare the time of vancomycin blood sample arrival at the lab after sampling in the control group versus intervention group

CONTACTS AND LOCATIONS:
Overall Officials: Birgit Koch, PharmD, Principal Investigator — Erasmus MC University Medical Center
Locations (1):
- Erasmus MC, Rotterdam, Netherlands